CLINICAL TRIAL: NCT00150670
Title: Randomized Phase III Study of TS-1 Alone Versus TS-1 Plus CDDP in Advanced Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Taiho Pharmaceutical Co., Ltd., Taiho Pharmaceutical Co., Ltd.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 91023039
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-07

CONDITIONS: Gastric Cancer
Keywords: Stomach cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — titanium silicide; Cisplatin

ARMS (2):
- 1 (Experimental): TS-1 and cisplatin
  Interventions: Drug: TS-1 and cisplatin
- 2 (Active Comparator): TS-1
  Interventions: Drug: TS-1

INTERVENTIONS:
Drug: TS-1 and cisplatin — TS-1(40-60 mg per body surface area) was given orally, twice daily for 3 consecutive weeks, and 60 mg/m2 cisplatin was given intravenously on day 8, followed by a 2-week rest period, within a 5-week cycle.
  Arms: 1
Drug: TS-1 — TS-1(40-60 mg per body surface area) was given orally, twice daily for 4 consecutive weeks, followed by a 2-week rest period, within a 6-week cycle.
  Arms: 2

SUMMARY:
This study aimed to verify the survival benefit of TS-1 plus CDDP combination chemotherapy compared with the monotherapy by TS-1 alone.

DETAILED DESCRIPTION:
This is a randomized, controlled, open-label, parallel, multicenter study. Patients are stratified according to 3 factors ; performance status (ECOG scale: 0, 1, 2), disease stage (unresectable gastric cancer or recurrent gastric cancer (received prior adjuvant chemotherapy or not)) and participating center. Patients are randomized to one of two treatment arms. Arm A: Patients receive oral TS-1 twice daily on days 1-28 followed by 14 days rest. Treatment is repeated every 42 days for up to 4 courses. Arm B: Patients receive CDDP iv on day 8 and oral TS-1 twice daily on days 1-21 followed by 14 days rest. Treatment is repeated every 35 days for up to 5 courses. Patients are followed every 6 months for up to 2 years from the day they participates in this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma
* Unresectable and recurrent gastric cancer
* Age 20 to 74
* Performance status 0, 1, or 2 (ECOG)
* Life expectancy 3 months
* No prior chemotherapy or radiotherapy for gastric cancer
* Able to take oral medication
* Evaluable or not evaluable lesion had already checked more than 28 days before participated in this study
* Hematopoietic Absolute granulocyte count lower limit of normal-12,000/mm^3 Platelet ≥ 100,000/mm^3 Hemoglobin ≥ 8.0 g/dL
* Hepatic AST and ALT ≤ 100 U/L ALP ≤ 2 times upper limit of normal (ULN) Bilirubin ≤ 1.5 mg/dL
* Renal Plasma creatinine ≤ ULN Creatinine clearance ≥ 50 mL/min

Exclusion Criteria:

* Pregnant or nursing
* Bleeding from gastrointestinal tract or no diarrhea
* Hypersensitivity to TS-1 or CDDP
* Psychiatric disorder that would preclude study compliance or giving informed consent
* Severe acute or chronic medical or psychiatric condition or laboratory abnormality
* Serious illness or medical condition
* Brain metastasis
* Ascites requiring drainage

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2002-03; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | every course for first three courses, then every other course

SECONDARY OUTCOMES:
Overall response rate, lesion-directed response rate, time to treatment failure (TTF), hospitalization-free survival period within the periods of TTF, and safety profile | every course for first three courses, then every other course

CONTACTS AND LOCATIONS:
Overall Officials: Wasaburo Koizumi, MD, PHD, Principal Investigator — East Hospital, Kitasato University
Locations (1):
- East Hospital, Kitasato University, 2-1-1, Asamizodai, Sagamihara, Kanagawa, Japan

REFERENCES:
- [Result] Koizumi W, Narahara H, Hara T, Takagane A, Akiya T, Takagi M, Miyashita K, Nishizaki T, Kobayashi O, Takiyama W, Toh Y, Nagaie T, Takagi S, Yamamura Y, Yanaoka K, Orita H, Takeuchi M. S-1 plus cisplatin versus S-1 alone for first-line treatment of advanced gastric cancer (SPIRITS trial): a phase III trial. Lancet Oncol. 2008 Mar;9(3):215-21. doi: 10.1016/S1470-2045(08)70035-4. Epub 2008 Feb 20. PMID 18282805
- [Derived] Arai H, Takeuchi M, Ichikawa W, Shitara K, Sunakawa Y, Oba K, Koizumi W, Sakata Y, Furukawa H, Yamada Y, Takeuchi M, Fujii M. Correlation of multiple endpoints in the first-line chemotherapy of advanced gastric cancer: Pooled analysis of individual patient data from Japanese Phase III trials. Cancer Med. 2024 Jan;13(1):e6818. doi: 10.1002/cam4.6818. Epub 2023 Dec 23. PMID 38140879